CLINICAL TRIAL: NCT00387543
Title: Review of Mayo Clinic Experience With Burning Mouth Syndrome - Use of Alpha Lipoic Acid
Brief Title: Alpha Lipoic Acid for Burning Mouth
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Other Study IDs: 06-002344
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Burning Sore Mouth

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Discussion and evaluation of patients with sore and burning mouth to determine whether alpha lipoic acid is helpful in managing their symptoms.

ELIGIBILITY:
Patients seen in the Department of Dermatology with diagnosis of burning mouth syndrome between 2000 and 2005

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: records of patients diagnosed with BMS in the Department of Dermatology between 1995 and 2005
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2000-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison J. Bruce, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States